CLINICAL TRIAL: NCT05429697
Title: Randomized, Placebo-controlled, Open-label, Phase 2b Clinical Trial to Evaluate the Antitumor Activity of Combination Therapy of SMT-NK and Pembrolizumab vs Pembrolizumab Monotherapy in Patients With Advanced Biliary Tract Cancer
Brief Title: Study of SMT-NK Inj. Plus Pembrolizumab vs Pembrolizumab Monotherapy in Patients With Advanced Biliary Tract Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: SMT bio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNK-SIT-03
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-06

CONDITIONS: Biliary Tract Cancer
Keywords: BTC; Cholangiocarcinoma; Biliary tract cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab+SMT-NK inj. (Experimental): Experimental:
  Pembrolizumab + SMT-NK inj. Participants will be randomized to receive 200 mg pembrolizumab followed by 3*10^6cells/kg SMT-NK inj.
  Interventions:
  Drug: SMT-NK inj. Drug: Pembrolizumab
  Interventions: Drug: SMT-NK inj.+Pembrolizumab
- Pembrolizumab (Placebo Comparator): Placebo Comparator: Pembrolizumb Participants will be randomized to receive 200 mg pembrolizumab.
  Intervention:
  Drug: Pembrolizumab
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: SMT-NK inj.+Pembrolizumab — SMT-NK inj. will be administered as an intravenous (IV) infusion on Day 1,Day 7 of each 21-day cycle.
  Pembrolizumab will be administered as an intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle.
  Arms: Pembrolizumab+SMT-NK inj.
Drug: Pembrolizumab — Pembrolizumab will be administered as an intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle.
  Arms: Pembrolizumab

SUMMARY:
This study is designed to assess the antitumor activity of combination therapy of SMT-NK (allogeneic natural killer cells) and pembrolizumab versus pembrolizumab monotherapy in patients with advanced biliary tract cancer

DETAILED DESCRIPTION:
The term of biliary tract cancer (BTC) refers to all tumors that arise from the biliary tract or the biliary drainage system, including the gallbladder.Biliary tract cancer is one of the most poorly prognosis cancers and the five-year survival rate remains at about 10% as it is difficult to expect long-term survival due to frequent local recurrence and remote metastasis after surgery.

South Korea belongs to a country with a high number of biliary tract cancer patients, and the incidence of biliary tract cancer is actually increasing every year.According to the 2018 National Cancer Registration Statistics, the number of 5-year biliary tract cancer patients was 13,967 (7,547 men and 6,420 women), which corresponds to about 2.9% of all cancersand the 5-year survival rate of biliary tract cancer patients between 2014 and 2018 was 28.8%, showing a lower survival rate than other cancer species.

Most of the long-term survival is due to early detection by screening, but advanced carcinoma is a refractory carcinoma with a 5-year survival rate of less than 5%.In addition to standard anticancer drugs, alternative anticancer drugs and targeted treatments can be developed for cancer with a large number of patients, but biliary tract cancer is difficult to find any more treatments if standard treatment fails and standard anticancer treatments cannot be continued due to resistance.

Natural killer cells (NK cells) are innate lymphocyte cells with cell killing activity, and have the characteristic of destroying cells by secretion of and granzyme into cancer cells and abnormal cells that are reduced or deficient in expression of MHC class I.Clinical studies using natural killer cells as anticancer drugs have long been conducted on various cancers.

Pembrolizumab is a monoclonal antibody designed to bind to a receptor called PD-1, which is expressed by immune cells such as T cells.Natural killer cells were also found to be expressing PD-1 in the same way as T cells, and in particular, PD-1 was found to be higher in cancer patients than in healthy people.

Therefore, combined therapy with the immune-check point such as pembrolizumab can be useful in elevating the anticancer activity of NK cells.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received a histopathological or cytologic diagnosis of nonresectable, advanced biliary tract carcinoma (intrahepatic or extrahepatic cholangiocarcinoma, gallbladder cancer) and patients with refractory disease after chemotherapy and/or patients who have difficulty with chemotherapy due to side effects of chemotherapy.
2. Patients who receives an explanation from the trial manager about the purpose, contents, and characteristics of the Investigational products for the clinical trial and is signed by the person, guardian or legal representative in the written informed consent.
3. 19 to 80 years old on day of signing informed consent.
4. Histopathological or cytologic diagnosis of advanced adenocarcinoma of the biliary tract and those with measurable lesions for RECIST evaluation

   * Tumor lesion: Must be accurately measured in at least one dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size of 10mm by CT scan
   * Malignant lymph nodes: To be considered pathologically enlarged and measurable, a lymph node must be ≥15mm in short axis when assessed by CT scan
5. Have a performance status of ≤2 on the ECOG Performance Scale.
6. Patients who survival period is expected to be at least 3 months.
7. Demonstrate laboratory test results the following conditions:

   * ANC (Absolute Neutrophil Count) ≥ 1,500/μL
   * Hemoglobin≥ 9 g/dL
   * Platelet> 80,000/μL
   * serum BUN & Creatinine ≤ 2.0 x upper limit of normal (ULN)
   * AST & ALT ≤ 5.0 x upper limit of normal (ULN)
   * Bilirubin ≤ 5mg/dL
   * Albumin ≥ 2.8g/dL
   * Prothrombin time (PT)% activity ≥ 70%
8. Patients or partners who has agreed to the appropriate use of contraceptives by two or more during the treatment period (including Survival follow-up period) (for men, those who have agreed not to provide sperm)
9. Patients who meet one or more of the following conditions:

   * Patients have at least 1% Combined Positive Score (*CPS) PD-L1 expression detected on the tumor, as determined by **immunohistochemistry performed by a central laboratory.

     * CPS = (number of PD-L1 positive tumor cells, lymphocytes, macrophage)/ (total number of viable tumor cells) X 100
     * Immunohistochemistry: IHC 22C3 pharmDx test

       ② Patients who have a positive MSI-H or dMMR test
       * MSI-high positive tumors analyzed by PCR
       * dMMR positive tumors analyzed by immunohistochemical staining
     * MSI-H was measured by PCR, and positive finding when two or more unstable markers were detected in PCR for 5 microsatellite markers, **dMMR is analyzed by immunohistochemical staining and positive when the discovery of one or more genes in MLH1, MSH2, MSH6 and PMS2 staining is lost.

Exclusion Criteria:

1. Patients who have previous history

   * Immune deficiency or autoimmune disease that can be aggravated by immunotherapy (for example: Rheumatoid arthritis, systemic lupus erythematosus, vasculitis, multiple sclerosis, Crohn's disease, ulcerative colitis, adolescent-developed insulin-dependent diabetes mellitus).
   * Immune deficiency disease
   * Pneumonia, colitis, hepatitis, nephritis, endocrine diseases associated with immunodeficiency (hypophysis, thyroid dysfunction, Type 1 diabetes, etc.)
   * Obvious myocardial failure or uncontrolled arterial hypertension
   * Active central nervous system (CNS) metastases and/or carcinomatous meningitis.
   * Non-infectious pneumonia, interstitial lung disease
   * Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
   * Hepatitis B (defined as HBsAg reactive) or known active hepatitis C virus (defined as HCV ribonucleic acid (RNA) [qualitative] is detected) infection or active tuberculosis
   * Active infection (if systemic treatment is required)
2. Has a diagnosed and/or treated additional malignancy within 5 years prior to signing informed consent except for curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin
3. Has a previous history of anti-angiogenic agent treatment before signing informed consent
4. Has a known serious allergic history
5. Has a known serious mental illness
6. Identified the following in Screening:

   * CRP ≥10 mg/dl and albumin ≤3.0 g/dl are suspected of cancer cachexia
   * Patients who have symptomatic ascites that is not controlled by medical treatment
7. Has received chemotherapy not less than 4 weeks old before randomization
8. Has received a live vaccine within 4 weeks before randomization
9. Is currently participating in or has participated in another clinical study within 4 weeks before randomization or the adverse event due to investigational drug administered remain before randomization
10. Has previously administrated Pembrolizumab and another anti-PD-1/PD-L1 agent
11. Has previously administrated immune-cell therapy (including natural killer cell etc.)
12. Female who are pregnant, breastfeeding or intending to become pregnant during the study period.
13. Has a history of any contraindication or has a severe hypersensitivity to any components of pembrolizumab
14. Has performed major surgery within 4 weeks prior to signing informed consent
15. Patients who are unsuitable to participate in clinical trials by investigator's decision

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2025-01-08 (Estimated); Study Completion 2026-06-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Up to approximately 72 weeks from the date of first administration of clinical trial drugs
  Progression-free survival (PFS) is defined as the time from the date of initial administration of the clinical trial drug to the progression or death due to any cause of the disease

SECONDARY OUTCOMES:
Object Response rate | Up to approximately 72 weeks from the date of first administration of clinical trial drugs
  Objective response rate (ORR) is defined as the ratio of subjects whose best overall response (hereinafter referred to as BOR) is partial response (PR) or complete response (CR) assessed by RECIST Version 1.1 and iRECIST.
Time to Progression | Up to approximately 72 weeks from the date of first administration of clinical trial drugs
  Time to disease progression (TTP) is defined as the time from the first administration date of the clinical trial drug to the first disease progression
Overall Survival | Up to approximately 120 weeks from the date of first administration of clinical trial drugs
  Overall survival(OS) is defined as the time from the date of first administration of the clinical trial drug to the death of all causes
Duration of Response | Up to approximately 72 weeks from the date of first administration of clinical trial drugs
  Duration of Response (DoR) is defined as the time from the date of the first documentation of objective response (confirmed CR or confirmed PR) to the date of the first disease progression or death due to any cause.
Disease Control Rate | Up to approximately 72 weeks from the date of first administration of clinical trial drugs
  Disease Control Rate (DCR) is defined as the proportion of participants who achieved a BOR of confirmed CR, confirmed PR, or stable disease (SD), assessed by RECIST Version 1.1 and iRECIST
Best Overall Response | Up to approximately 72 weeks from the date of first administration of clinical trial drugs
  In order for the best overall response (BOR) to be finally evaluated as partial response (PR) or complete response (CR), it must be evaluated as partial response (PR) or complete response (CR) in two consecutive evaluations by RECIST Version 1.1 and iRECIST.
Time to Response | Up to approximately 72 weeks from the date of first administration of clinical trial drugs
  The time to response (TTR) is defined as the time from the date of first administration of the clinical trial drug to the time when it is evaluated as the first partial response (PR) or full response (CR) by RECIST Version 1.1 and iRECIST.
Quality of Life | Up to approximately 72 weeks from the date of first administration of clinical trial drugs
  Assessed by EORTC-QLQ(The European Organization for Research and Treatment-QoL questionnaire) C30

CONTACTS AND LOCATIONS:
Overall Officials: SEUNGWOO PARK, Principal Investigator — Department of Internal Medicine, Yonsei University College of Medicine, Severance Hospital
Locations (3):
- South Korea (3):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Severance Hospital, Seoul
  - Gangnam Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No